CLINICAL TRIAL: NCT05604417
Title: A Phase 1 Study With a Phase 2 Expansion Cohort of Zandelisib and Tazemetostat in Relapsed or Refractory Follicular Lymphoma
Brief Title: Zandelisib + Tazemetostat in R/R Follicular Lymphoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Termination of Zandelisib clinical development globally
Sponsor: Jacob Soumerai, MD (Other)
Collaborators: MEI Pharma, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Jacob Soumerai, MD, Sponsor Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-103
Record Dates: First submitted 2022-10-28; First posted 2022-11-03 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Relapsed Follicular Lymphoma; Refractory Follicular Lymphoma
Keywords: Relapsed Follicular Lymphoma; Refractory Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — tazemetostat; ME-401

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PHASE 1: ZANDELISIB + TAZEMETOSTAT (Experimental): Phase 1 study (3+3 design), followed by a phase 2 expansion component
  * For phase 1 portion, which follows the same dosing schedule as Arm A, there will not be any randomization.
  * Zandelisib, oral, daily on predetermined days each cycle for a total of 14 cycles
  * Tazemetostat oral, twice daily on predetermined days (Cycles 1) and predetermined days (Cycles 2-14) for a total of 14 cycles. There will be 2 dose levels of tazemetostat.
  Interventions: Drug: TAZEMETOSTAT; Drug: Zandelisib
- Arm A: COMBINATION ZANDELISIB + TAZEMETOSTAT (Experimental): Participants randomized into Arm A of the phase 2 component will receive
  * Zandelisib, oral, daily on predetermined days each cycle for a total of 14 cycles
  * Tazemetostat oral, twice daily on predetermined days (Cycles 1) and predetermined days (Cycles 2-14) for a total of 14 cycles
  Interventions: Drug: TAZEMETOSTAT; Drug: Zandelisib
- Arm B: Zandelisib and Tazemetostat (Experimental): Participants randomized into Arm B of the phase 2 component will receive
  * Zandelisib oral, daily on predetermined days (Cycles 1-2) and predetermined days of cycle 3 and onwards up to 14 cycles.
  * Tazemetostat, oral, twice daily on predetermined days of each cycle. This will begin on cycle 3 and will continue for up to 12 cycles.
  Interventions: Drug: TAZEMETOSTAT; Drug: Zandelisib

INTERVENTIONS:
Drug: TAZEMETOSTAT — Dosage and treatment timings per protocol
  Other Names: TAZVERIK
Drug: Zandelisib — Dosage and treatment timings per protocol
  Other Names: ME-401

SUMMARY:
This research study is being done to estimate the safety and efficacy of zandelisib and tazemetostat in people with relapsed or refractory follicular lymphoma (FL)

This research study involves Zandelisib in combination with Tazemetostat.

MEI Pharma, Inc, a biotechnology company, is supporting this research study by providing funding for the research study, including the study drug zandelisib.

DETAILED DESCRIPTION:
This is a phase 1 study of Zandelisib and Tazemetostat with a phase 2 expansion two-arm component in patients with relapsed or refractory follicular lymphoma (FL) grade 1-3A.

- This research study involves Zandelisib in combination with Tazemetostat. This is the first time the drug combination of Zandelisib and Tazemetostat will be given to humans.

* The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits
* Participants will receive study treatment as long as treatment is tolerated and the disease does not worsen.
* The maximum length of time on the study drug combination is 14 months. Participants will followed for up to 2 years.
* It is expected that about 34 people will take part in this research study.

The U.S. Food and Drug Administration (FDA) has not approved zandelisib as a treatment for any disease.

The U.S. FDA has approved tazemetostat as a treatment for relapsed or refractory follicular lymphoma as a single therapy.

This is the first time this drug combination will be given to humans. This is a Phase I/II clinical trial. Participants will be asked to participate in either the Phase I part or Phase II part of this clinical trial.

* A Phase I clinical trial tests the safety of an investigational drug and also tries to define the appropriate dose of the investigational drug to use for further studies.
* A Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease.

"Investigational" means that the drug is being studied.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have biopsy-proven relapsed or refractory FL grade 1-2 or 3A by WHO criteria.
* Participants must require therapy based on: symptomatic disease, threatened end-organ dysfunction, compressive disease, cytopenias secondary to lymphoma, bulky disease (defined as any site 7 cm or greater in size, or 3 or more sites 3 cm or greater in size), or progression.
* Participants must have received at least two prior systemic therapies for FL, or have relapsed or refractory FL who have no satisfactory alternative treatment options.
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of zandelisib in combination with tazemetostat in participants <18 years of age, children are excluded from this study.
* ECOG performance status ≤2 (Karnofsky ≥60%).
* Participants must have adequate marrow function as defined below (unless abnormalities are considered related to marrow and/or splenic involvement by lymphoma):

  * absolute neutrophil count ≥1,000/mcL
  * platelets ≥75,000/mcL
* Participants must have adequate organ function as defined below (unless abnormalities are considered related to target organ involvement or compression by lymphoma):

  * total bilirubin ≤ 1.5x institutional upper limit of normal (ULN) (Isolated bilirubin ≤3.0x ULN is acceptable if considered secondary to Gilbert's syndrome)
  * AST(SGOT)/ALT(SGPT) ≤2.0 × institutional ULN Creatinine clearance ≥50 mL/min eGFR (Cockcroft-Gault)
* Participants with known history or current symptoms of cardiac disease should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* The effects of zandelisib and tazemetostat on the developing human fetus are unknown. A female participant is eligible to participate if she is not pregnant or breastfeeding. Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, and for at least 4 months after the last dose of study intervention. Women must also agree not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Nonchildbearing potential is defined as follows (by other than medical reasons):

  * ≥45 years of age and has not had menses for >1 year
  * Patients who have been amenorrhoeic for <1 year without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
  * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure.
* Women of childbearing potential must have a negative highly sensitive serum pregnancy test, and agree to repeat the highly sensitive serum pregnancy testing within 72 hours before the first dose of study intervention (if screening pregnancy test was not within 72 hours of dosing).
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of administration. Men must also agree not to donate sperm during this period. Men may agree to remain abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term or persistent basis) OR agree to use a male condom, even if they have undergone a successful vasectomy and female partner to use an additional highly effective contraceptive method with a failure rate of <1% per year when having sexual intercourse with a WOCBP (including pregnant females).
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia. At the discretion of the overall PI, participants with residual toxicities >Grade 1 may be considered eligible if in the opinion of the overall PI the residual toxicity is not likely to interfere with the safety or efficacy assessment of the investigational regimen.
* Participants who are receiving any other investigational agents.
* Participants must not have known central nervous system involvement by lymphoma.
* Participant must not have used an investigational drug or approved systemic lymphoma therapy with 14 days or five half-lives, whichever is shorter, preceding the first dose of study drug. Steroids are permitted.
* Participant must not have received a PI3K inhibitor or EZH2 inhibitor.
* Participants must not have known immediate or delayed hypersensitivity reaction or idiosyncratic reactions to zandelisib, tazemetostat, or drugs chemically related to zandelisib or tazemetostat, or any of the components of the study treatment.
* Participants must not have an uncontrolled intercurrent illness.
* Participants must not have an uncontrolled active infection.
* Participants must not have inflammatory bowel disease.
* Participants must not have active uncontrolled autoimmune disease.
* Participants must not have psychiatric illness/social situations that would limit compliance with study requirements. Participants must not have any serious and/or preexisting medical or other condition (including lab abnormalities) that could interfere with participant's safety in the opinion of the investigator.
* Women who are pregnant are excluded from this study because it is unknown if tazemetostat or zandelisib can cause embryo-fetal harm when administered to a pregnant woman. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with zandelisib and tazemetostat, breastfeeding should be discontinued if the mother is treated with zandelisib and tazemetostat.
* Participants must not have an active malignancy or systemic therapy for another malignancy within 3 years; local/regional therapy with curative intent such as surgical resection or localized radiation within 3 years of treatment is permitted; active prostate cancer that is considered low-risk and appropriate for continued active surveillance strategy is permitted. Additionally, adequately treated basal, squamous cell carcinoma, or non-melanomatous skin cancer, carcinoma in situ of the cervix, or superficial bladder cancer not treated with intravesical chemotherapy or BCG within 6 months, are permitted.
* Participant must be able to swallow pills.
* Participant must not have active uncontrolled HIV infection. Participants with HIV are eligible if disease is adequately controlled, defined by presence of both an undetectable viral load and a CD4 count >200.
* Participant must not have active hepatitis B infection. Participant with positive HBV core antibody or HBV surface antigen at screening are eligible if HBV viral load is negative by PCR and on appropriate antiviral therapy. Participant must not have active hepatitis C infection. Note: participants with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C RNA test is obtained. Note: Hepatitis RNA testing is optional and participants with negative Hepatitis C antibody test are not required to also undergo Hepatitis C RNA testing.
* Coadministration of strong or moderate CYP3A inhibitors or inducers is not permitted. If a patient is taking a strong or moderate CYP3A inhibitor or inducer prior to starting treatment, this medication needs to be stopped for 1 week prior to initiation of protocol therapy to allow for a washout period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities Phase I | Up to 28 days
  Dose-limiting toxicity (DLT) is defined as an Adverse Event (AE) that meets all of the following criteria: Occurs during the 28 days of cycle 1 (DLT window); Is deemed at least possibly related to protocol therapy
Complete Response Rate Phase II | up to 4 years
  response classified per the 2014 Lugano criteria

SECONDARY OUTCOMES:
Overall Response Rate | Up to 4 years
  Response classified per the 2014 Lugano criteria
Median Progression-Free Survival | as the time from registration to the earlier of progression or death due to any cause up to 4 years
  summarized using Kaplan-Meier method
Overall Survival | as the time from registration to death due to any cause, or censored at date last known alive up to 4 years
  summarized using Kaplan-Meier method
Duration of Response | Up to 4 years
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented summarized using Kaplan-Meier method
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | baseline up to 4 years
  NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jacob D. Soumerai, MD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation